CLINICAL TRIAL: NCT01222052
Title: Randomized Multicenter Study Comparing 6xFEC With 3xFEC-3xDoc in High-risk Node-negative Patients With Operable Breast Cancer: Comparison of Efficacy and Evaluation of Clinico-pathological and Biochemical Markers as Risk Selection Criteria
Brief Title: 6xFU/Epirubicin/Cyclophosphamide (FEC) Compared to 3xFEC-3xDocetaxel in High-risk Node-negative Breast Cancer Patients
Acronym: NNBC3-Europe
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Collaborators: GBG Forschungs GmbH (Other)
Responsible Party: Principal Investigator, Christoph Thomssen, Prof. Dr. Christoph Thomssen, Martin-Luther-Universität Halle-Wittenberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBG 42; NCT02681003 (obsolete NCT alias)
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer
Keywords: high risk breast cancer; low risk breast cancer; uPA; urokinase-type plasminogen activator; PAI; plasminogen activator inhibitor-type
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; Epirubicin; Cyclophosphamide; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A Taxane-containing (Experimental): 3 courses FEC q3weeks followed by 3 courses Docetaxel q3weeks
  Interventions: Drug: 5-Fluorouracil, Epirubicin, Cyclophosphamide, Docetaxel
- Arm B standard anthracyclin (Active Comparator): 6 courses of FEC q3weeks
  Interventions: Drug: 5-Fluorouracil, Epirubicin, Cyclophosphamide, Docetaxel
- Observation (No Intervention)

INTERVENTIONS:
Drug: 5-Fluorouracil, Epirubicin, Cyclophosphamide, Docetaxel — Arm A 5-FU 500mg/m2, Epirubicin 100mg/m2, Cyclophosphamide 500mg/m2 q3weeks followed by Docetaxel 100 mg/m² q3weeks
  Arm B 5-FU 500mg/m2, Epirubicin 100mg/m2, Cyclophosphamide 500mg/m2 q6weeks
  Arms: Arm A Taxane-containing; Arm B standard anthracyclin

SUMMARY:
In low-risk node-negative breast cancer patients adjuvant chemotherapy should be spared. The identification of this subgroup can be based either on clinical and pathological or on tumour-biological criteria. Due to their high prognostic impact, the tumour-biological invasion markers uPA/PAI-1 (urokinase-type plasminogen activator and its inhibitor PAI-1) are potential candidates to effectively assess the risk of relapse in node-negative breast cancer. This study is aimed to compare the risk assessment by the traditional clinico-pathological factors and by tumour-biological factors. The second study question refers to the comparison between an adjuvant combination treatment with FE100C*6 and a sequential treatment with FE100C*3 and Docetaxel*3.

DETAILED DESCRIPTION:
1. To compare FEC*6 with FEC*3 followed by DOC*3 with regard to:

   * the primary endpoint of the study: Disease-Free Survival (DFS)
   * the secondary endpoints: Overall Survival (OS), compliance, and toxicity of chemotherapy in each patient group
2. To compare patients with low risk according to clinico-pathological versus those according to biological risk criteria with regard to:

   * the proportion of low risk versus high risk patients
   * DFS
   * OS (secondary endpoint)

ELIGIBILITY:
Inclusion Criteria:

* Histological proven primary breast cancer
* Tumour size >0.5 cm and <5 cm (pT1b-pT2, pN0, M0)
* Axillary lymph nodes tumour free (node-negative disease)
* Adequate surgical procedure: R0-resection and axillary dissection with more than 10 lymph nodes examined or adequate sentinel procedure in a qualified centre
* Frozen tumour tissue available (for analysis of biological markers and microarrays, centres with biological risk assessment only). The material has to be stored in liquid nitrogen immediately after excision.
* Paraffin blocks or (at least) pathology slides of primary tumour (stained and unstained) and axillary nodes (stained) available for central review.
* HER-2/neu determination by immunohistochemistry. Patients will be stratified to be HER-2/neu-negative or HER-2/neu-positive (HER-2/neu Score 3+, or HER-2/neu Score 2+ and FISH positive).
* No distant metastasis
* Age >18 years, <70 years
* Performance status ECOG <2 (WHO Performance Status 0-1)
* Adequate cardiac function (echocardiographically measured left ventricular ejection fraction (LVEF) or shortening fraction (SF) within the normal limits, i.e. ≥55%)
* Adequate bone function (neutrophil count >1.5 x109 /l and platelet count >100 x109 /l)
* Adequate renal function (serum creatinine <120 µmol/l or 1.35 mg/dl) and hepatic function (serum bilirubin <1 x UNL, ASAT or ALAT (SGOT or SGPT) <2,5 x UNL)
* Before patient registration/randomization, written informed consent must be obtained according to ICH/EU GCP, and national/local regulations

Exclusion Criteria:

* Chemotherapy contraindicated
* Inflammatory breast cancer, tumour infiltrated axillary lymph nodes including the sentinel node.
* Other concomitant pathology compromising survival (at entry), or preventing the administration of chemotherapy with either FEC or Docetaxel
* Other serious illness or medical condition that may interfere with the understanding and giving of informed consent and the conduct of the study
* Estimated life-expectancy <10 years (irrespective of breast cancer diagnosis)
* Patient not accessible for treatment and follow up
* Endocrine treatment not according to the latest standard recommendations of the AGO Kommission "Mamma"
* Pregnancy, lactation (sufficient non-hormonal contraception in fertile women required)
* Surgery more than six weeks ago at the start of chemotherapy
* Pre-existing polyneuropathy
* Previous or concomitant other malignancy (including contralateral breast cancer) except adequately treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix
* Prior chemotherapy or radiotherapy or endocrine therapy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4150 (Actual)
Dates: Start 2002-01; Primary Completion 2009-02 (Actual); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival | after 10 years follow up

SECONDARY OUTCOMES:
Overall Survival | after 10 years follow up

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Thomssen, MD, Principal Investigator — Dpt. Gynecology University Halle Germany; Nadia Harbeck, MD, Principal Investigator — Breast Center University Cologne
Locations (1):
- GBG Forschungs GmbH, Neu-Isenburg, Germany

REFERENCES:
- [Derived] Kantelhardt EJ, Vetter M, Schmidt M, Veyret C, Augustin D, Hanf V, Meisner C, Paepke D, Schmitt M, Sweep F, von Minckwitz G, Martin PM, Jaenicke F, Thomssen C, Harbeck N. Prospective evaluation of prognostic factors uPA/PAI-1 in node-negative breast cancer: phase III NNBC3-Europe trial (AGO, GBG, EORTC-PBG) comparing 6xFEC versus 3xFEC/3xDocetaxel. BMC Cancer. 2011 Apr 16;11:140. doi: 10.1186/1471-2407-11-140. PMID 21496284